CLINICAL TRIAL: NCT01159535
Title: Mindfulness Based Relapse Prevention: Efficacy and Mechanisms
Acronym: MBRP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Seema Clifasefi, Assistant Professor/Co-Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 31183-J; 1R01DA025764-01A1 (NIH)
Record Dates: First submitted 2010-07-07; First posted 2010-07-09 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-07

CONDITIONS: Substance Use Disorders
Keywords: substance use; addiction; meditation; mindfulness; relapse prevention
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive | interventions — Secondary Prevention; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MBRP (Active Comparator): The Mindfulness Based Relapse Prevention (MBRP) intervention is composed of 8 weekly 2-hour sessions delivered in small group format (10-14 participants). Individual sessions will be team-taught by two therapists and will include mindfulness practices targeting craving, Negative affect, and reactivity, as well as discussion about how to implement practice into high-risk situations and in daily life.
  Interventions: Behavioral: Mindfulness Based Relapse Prevention
- Relapse Prevention (RP) (Active Comparator): The RP intervention is composed of 8 weekly 2-hour sessions delivered in small group format (10-14 participants). Individual sessions will be team-taught by two therapists and will include discussions of personal high-risk situations, coping skills assessment, and exercises to evaluate expectancies, self-efficacy, and craving.
  Interventions: Behavioral: Relapse Prevention
- Treatment as Usual (Active Comparator): All participants will be enrolled in continuing care services (including attendance at AA, NA, or other self-help groups) as recommended by their treatment providers. Thus, TAU participants will have ongoing support and monitoring by their continuing care providers on a regular basis.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Mindfulness Based Relapse Prevention — The MBRP intervention comprises 8 weekly, 2-hour sessions delivered in small group format (10-14 participants) by two therapists (Bowen, et al., 2009). In MBRP, therapists facilitate discussions and exercises and introduce the meditation practice component.Group sessions include discussions of mindfulness as a means of coping with craving and painful cognitions/sensations that precipitate relapse, role-playing exercises, meditation practice, and homework assignments.
  Other Names: MBRP
  Arms: MBRP
Behavioral: Relapse Prevention — intervention is composed of 8 weekly 2-hour sessions delivered in small group format (10-14 participants)
  Other Names: RP
  Arms: Relapse Prevention (RP)
Behavioral: Treatment as Usual — All participants will be enrolled in continuing care services (including attendance at AA, NA, or other self-help groups) as recommended by their treatment providers. Thus, TAU participants will have ongoing support and monitoring by their continuing care providers on a regular basis.
  Other Names: TAU
  Arms: Treatment as Usual

SUMMARY:
The broad, long-term objective of the proposed randomized clinical trial is to evaluate the efficacy, moderators and mechanisms of change of two cognitive-behavioral aftercare treatments for alcohol and other drug (AOD) use disorders in preventing AOD relapse compared to treatment as usual (TAU) offered in the community. The two cognitive-behavioral aftercare treatments are relapse prevention (RP) and Mindfulness-Based Relapse Prevention (MBRP), which integrates mindfulness meditation and RP aftercare components.

DETAILED DESCRIPTION:
Relapse to alcohol and other drug use (AOD) following treatment continues to be a costly problem for individual, society, and the substance abuse treatment community, and thus warrants the continued development of innovative and efficacious interventions designed to prevent AOD relapse. Mindfulness based relapse prevention (MBRP; Bowen, Chawla, & Marlatt, 2008) is one such promising intervention: it incorporates mindfulness meditation on the foundation of cognitive-behavioral relapse prevention (RP;Daley & Marlatt, 2006). RP is an established substance abuse treatment, yet as treatment developers, we believe RP can continue to be enhanced. Based on the results of an initial pilot trial, MBRP has demonstrated both feasibility and empirical promise as an aftercare treatment for AOD disorders in further enhancing long-term behavior change and reducing risk of relapse and related consequences. In the proposed study, MBRP and RP will be compared to the treatment as usual (TAU) as delivered by the Recovery Centers of King County (RCKC), in a population of individuals who have received community-based intensive inpatient (IP) or outpatient (IOP) treatment. RCKC is a community treatment agency that provides a range of addiction treatment services and has previously supported our efforts to recruit and retain sufficient numbers of the target population. The proposed study will examine whether structured mindfulness practice results in fewer AOD use days and fewer problems related to AOD use compared to TAU over a longer-term followup than in the previous pilot study. Given the high prevalence of AOD abuse in the population and the high rates of relapse following AOD treatment, the proposed research will provide a valuable next step in evaluating the efficacy of MBRP as an aftercare treatment for AOD disorders and in understanding the mechanisms of treatment efficacy. To our knowledge, no prior substance abuse treatment studies have evaluated the effect of adding a mindfulness-based component (e.g., MBRP) to an existing empirically supported treatment (i.e., RP).

ELIGIBILITY:
Inclusion Criteria:

* completion or scheduled completion (i.e., within 2 weeks) of Inpatient or Intensive Outpatient treatment
* fluency in English
* enrollment in a substance abuse aftercare program
* medical clearance by referring provider
* willingness to accept random assignment to treatment condition

Exclusion Criteria:

* already participated in the pilot MBRP trial conducted by this research team
* participation in the comorbid disorders or relapse prevention groups offered at partner agency
* comorbid psychosis (including schizophrenia, schizoaffective or other schizophreniform disorder)and/or dementia, acute suicidality/intent to harm others, severe cognitive impairment, and high risk of withdrawal or medical complications stemming from relapse which would require a higher level of care.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2009-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Bowen, PhD, Principal Investigator — University of Washington
Locations (1):
- Recovery Centers of King County, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bowen S, Chawla N, Collins SE, Witkiewitz K, Hsu S, Grow J, Clifasefi S, Garner M, Douglass A, Larimer ME, Marlatt A. Mindfulness-based relapse prevention for substance use disorders: a pilot efficacy trial. Subst Abus. 2009 Oct-Dec;30(4):295-305. doi: 10.1080/08897070903250084. PMID 19904665
- [Background] Witkiewitz K, Bowen S. Depression, craving, and substance use following a randomized trial of mindfulness-based relapse prevention. J Consult Clin Psychol. 2010 Jun;78(3):362-374. doi: 10.1037/a0019172. PMID 20515211
- [Background] Bowen S, Witkiewitz K, Dillworth TM, Marlatt GA. The role of thought suppression in the relationship between mindfulness meditation and alcohol use. Addict Behav. 2007 Oct;32(10):2324-8. doi: 10.1016/j.addbeh.2007.01.025. Epub 2007 Jan 23. PMID 17300875
- [Background] Bowen S, Witkiewitz K, Dillworth TM, Chawla N, Simpson TL, Ostafin BD, Larimer ME, Blume AW, Parks GA, Marlatt GA. Mindfulness meditation and substance use in an incarcerated population. Psychol Addict Behav. 2006 Sep;20(3):343-7. doi: 10.1037/0893-164X.20.3.343. PMID 16938074
- [Background] Chawla N, Collin S, Bowen S, Hsu S, Grow J, Douglass A, Marlatt GA. The mindfulness-based relapse prevention adherence and competence scale: development, interrater reliability, and validity. Psychother Res. 2010 Jul;20(4):388-97. doi: 10.1080/10503300903544257. PMID 20204916
- [Background] Collins SE, Chawla N, Hsu SH, Grow J, Otto JM, Marlatt GA. Language-based measures of mindfulness: initial validity and clinical utility. Psychol Addict Behav. 2009 Dec;23(4):743-9. doi: 10.1037/a0017579. PMID 20025383
- [Derived] Somohano VC, Rehder KL, Dingle T, Shank T, Bowen S. PTSD Symptom Clusters and Craving Differs by Primary Drug of Choice. J Dual Diagn. 2019 Oct-Dec;15(4):233-242. doi: 10.1080/15504263.2019.1637039. Epub 2019 Jul 14. PMID 31304887
- [Derived] Bowen S, Witkiewitz K, Clifasefi SL, Grow J, Chawla N, Hsu SH, Carroll HA, Harrop E, Collins SE, Lustyk MK, Larimer ME. Relative efficacy of mindfulness-based relapse prevention, standard relapse prevention, and treatment as usual for substance use disorders: a randomized clinical trial. JAMA Psychiatry. 2014 May;71(5):547-56. doi: 10.1001/jamapsychiatry.2013.4546. PMID 24647726

RESULTS

PARTICIPANT FLOW:
Groups:
- Mindfulness Based Relapse Prevention (MBRP): Mindfulness Based Relapse Prevention
  Mindfulness Based Relapse Prevention: The MBRP intervention comprises 8 weekly, 2-hour sessions delivered in small group format (10-14 participants) by two therapists (Bowen, et al., 2009). In MBRP, therapists facilitate discussions and exercises and introduce the meditation practice component.Group sessions include discussions of mindfulness as a means of coping with craving and painful cognitions/sensations that precipitate relapse, role-playing exercises, meditation practice, and homework assignments.
- Treatment as Usual (TAU): All participants will be enrolled in continuing care services (including attendance at AA, NA, or other self-help groups) as recommended by their treatment providers. Thus, TAU participants will have ongoing support and monitoring by their continuing care providers on a regular basis.
  Treatment as Usual: All participants will be enrolled in continuing care services (including attendance at AA, NA, or other self-help groups) as recommended by their treatment providers. Thus, TAU participants will have ongoing support and monitoring by their continuing care providers on a regular basis.
Period: Overall Study
Arm/Group | Mindfulness Based Relapse Prevention (MBRP) | Relapse Prevention (RP) | Treatment as Usual (TAU)
Started | 103 | 88 | 95
Completed | 79 | 64 | 64
Not Completed | 24 | 24 | 31

BASELINE CHARACTERISTICS:
Groups:
- Mindfulness Based Relapse Prevention (MBRP): Mindfulness Based Relapse Prevention: The MBRP intervention comprises 8 weekly, 2-hour sessions delivered in small group format (10-14 participants) by two therapists (Bowen, et al., 2009). In MBRP, therapists facilitate discussions and exercises and introduce the meditation practice component.Group sessions include discussions of mindfulness as a means of coping with craving and painful cognitions/sensations that precipitate relapse, role-playing exercises, meditation practice, and homework assignments.
- Total: Total of all reporting groups
Arm/Group | Mindfulness Based Relapse Prevention (MBRP) | Relapse Prevention (RP) | Treatment as Usual | Total
Number analyzed (Participants) | 103 | 88 | 95 | 286
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 103 | 88 | 95 | 286
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (10.9) | 38.9 (10.9) | 37.2 (10.8) | 38.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 32 | 26 | 85
  Male | 76 | 56 | 69 | 201
Region of Enrollment [Number; unit: participants]
  United States | 103 | 88 | 95 | 286

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Alcohol and Drug Use Days Out of Past 30
Description: Self reported use of alcohol and or illicit substances over the previous 30 days
Time Frame: 30 days previous, assessed at 12-month follow-up
Measure: Mean (Standard Deviation); unit: number of days out of past 30
Groups:
- Mindfulness Based Relapse Prevention (MBRP): Mindfulness Based Relapse Prevention
  Mindfulness Based Relapse Prevention: The MBRP intervention consisted of 8 weekly, 2-hour sessions delivered in small group format (10-14 participants) by two therapists (Bowen, et al., 2009). In MBRP, therapists facilitate discussions and exercises and introduce the meditation practice component.Group sessions include discussions of mindfulness as a means of coping with craving and painful cognitions/sensations that precipitate relapse, role-playing exercises, meditation practice, and homework assignments.
- Treatment as Usual (TAU): Treatment as Usual included continuing care services (including attendance at Alcoholics Anonymous, Narcotics Anonymous, or other self-help groups) as recommended by their treatment providers.
Arm/Group | Mindfulness Based Relapse Prevention (MBRP) | Relapse Prevention (RP) | Treatment as Usual (TAU)
Number analyzed (Participants) | 103 | 88 | 95
number of days out of past 30
  Mean number of heavy drinking days | 1.44 (7.66) | 3.89 (12.17) | 4.65 (14.93)
  Mean number of drug use days | 3.06 (15.08) | 6.09 (19.05) | 4.63 (16.03)

ADVERSE EVENTS:
Groups:
- Mindfulness-Based Relapse Prevention (MBRP): Mindfulness Based Relapse Prevention comprises 8 weekly, 2-hour sessions delivered in small group format (10-14 participants) by two therapists (Bowen, et al., 2009). In MBRP, therapists facilitate discussions and exercises and introduce the meditation practice component.Group sessions include discussions of mindfulness as a means of coping with craving and painful cognitions/sensations that precipitate relapse, role-playing exercises, meditation practice, and homework assignments.
- Relapse Prevention (RP): The RP intervention is composed of 8 weekly 2-hour sessions delivered in small group format (10-14 participants). Individual sessions were team-taught by two therapists and will include discussions of personal high-risk situations, coping skills assessment, and exercises to evaluate expectancies, self-efficacy, and craving.
  Relapse Prevention: intervention is composed of 8 weekly 2-hour sessions delivered in small group format (10-14 participants)
- Treatment as Usual (TAU): Treatment as Usual participants were enrolled in continuing care services (including attendance at AA, NA, or other self-help groups) as recommended by their treatment providers. Thus, TAU participants received ongoing support and monitoring by their continuing care providers on a regular basis.
Arm/Group | Mindfulness-Based Relapse Prevention (MBRP) | Relapse Prevention (RP) | Treatment as Usual (TAU)
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/88 | 0/95
Other Adverse Events (participants affected / at risk) | 0/103 | 0/88 | 0/95

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes